CLINICAL TRIAL: NCT04265430
Title: Serial Magnetic Resonance Imaging of Longitudinal Radiotherapy-Attributable Normal Tissue Injury
Brief Title: Serial Magnetic Resonance Imaging for the Prediction of Radiation-Induced Changes in Normal Tissue of Patients With Oral Cavity or Skull Base Tumors
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PA14-0807; NCI-2019-07862 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PA14-0807 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-12-03; First posted 2020-02-11 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Malignant Oral Cavity Neoplasm; Malignant Skull Base Neoplasm; Osteoradionecrosis
MeSH Terms: conditions — Mouth Neoplasms; Osteoradionecrosis | interventions — Contrast Media; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort I (MRI after radiation therapy) (Experimental): Patients may receive a contrast agent IV and then undergo an MRI over 45-60 minutes at baseline, 3-5 weeks after starting standard of care radiation therapy, and then at 2 months, 6 months, 12 months, and 3 years after completing radiation therapy.
  Interventions: Other: Contrast Agent; Procedure: Magnetic Resonance Imaging; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Cohort II (MRI after surgery) (Experimental): Patients may receive a contrast agent IV and then undergo an MRI over 45-60 minutes at baseline, and at 5-10 weeks and 12 months after standard of care surgery.
  Interventions: Other: Contrast Agent; Procedure: Magnetic Resonance Imaging; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Contrast Agent — Given IV
  Other Names: Contrast; Contrast Drugs; contrast material; Contrast Medium
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase IV trial studies how well serial magnetic resonance imaging (MRI) after radiation therapy works in predicting radiation-induced changes in the normal tissue of patients with oral cavity or skull base tumors. Performing MRIs after radiation therapy for patients with oral cavity or skull base tumors may help to predict osteoradionecrosis (a change in non-cancerous tissue).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Demonstrate the feasibility of serial magnetic resonance (MR) imaging biomarkers for assessment of early, intermediate, and late radiotherapy-attributable physiologic alteration of tumor and normal tissues and the kinetics thereof.

II. Develop MR-biomarker inclusive predictive models for development of radiotherapy-attributable normal tissue injury.

III. Define dose-response relationships between imaging biomarkers and subsequent radiation-induced effects.

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHORT I: Patients may receive a contrast agent intravenously (IV) and then undergo an MRI over 45-60 minutes at baseline, 3-5 weeks after starting standard of care radiation therapy, and then at 2 months, 6 months, 12 months, and 3 years after completing radiation therapy.

COHORT II: Patients may receive a contrast agent IV and then undergo an MRI over 45-60 minutes at baseline, and at 5-10 weeks and 12 months after standard of care surgery.

ELIGIBILITY:
Inclusion Criteria:

All Cohorts:

* Patients older than 18 years of age
* Patients with good performance status (ECOG score 0-2)
* Patients willing to give written informed consent.

Cohort 1 (Individuals without ORN or MRONJ):

* Patients with histologically proven malignant neoplasms of the oral cavity, oropharynx or skull base.
* Patients currently dispositioned to treatment with radiotherapy and/or antiresorptive or antiangiogenic medication therapy

Cohort 2 (Individuals with ORN or MRONJ):

* Patients with a clinical diagnosis of ORN or MRONJ following treatment for cancer
* Patients previously dispositioned to treatment with radiotherapy and/or antiresorptive or antiangiogenic medication therapy

Exclusion Criteria:

* Patients unable to tolerate DW-MRI or DCE-MRI or having an estimated GFR < 30ml/min/1.73m2.
* Patients with contraindication to MRI (e.g. non-MRI compatible metallic implants)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 425 (Estimated)
Dates: Start 2018-09-17 (Actual); Primary Completion 2031-09-01 (Estimated); Study Completion 2031-09-01 (Estimated)

PRIMARY OUTCOMES:
Radiotherapy-attributable imaging for normal tissue injury | Up to 1 year
  Will correlate whether post-therapy alterations in the observed multi-parametric imaging features can be used as surrogate bio-markers of normal tissue injury
Dose-response correlation between imaging biomarkers | Up to 1 year
  Penalized spline mixed regression will be used to characterize the induced functional relationships between the delivered dose and imaging biomarkers identified at each imaging time point. Doses for which 95% confidence interval estimates of mean trajectory fail to overlap will characterize ranges that yield significantly different levels of dose-dependent modulation.
Dose-response correlation between subsequent radiation-induced effects | Up to 1 year
  Penalized spline mixed regression will be used to characterize the induced functional relationships between the delivered dose and imaging biomarkers identified at each imaging time point. Doses for which 95% confidence interval estimates of mean trajectory fail to overlap will characterize ranges that yield significantly different levels of dosedependent modulation

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Y Lai, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org